CLINICAL TRIAL: NCT06253169
Title: Benefit of Self-sampling for HPV DNA in a General Practitioner's Office to Improve Participation in Cervical Screening - The ASTRA Study.
Brief Title: HPV DNA Self-sampling in a General Practitioner's Office.
Acronym: ASTRA
Status: Recruiting | Type: Observational
Sponsor: Patient Organization Veronica (Other Government)
Responsible Party: Sponsor
Other Study IDs: V01
Record Dates: First submitted 2024-01-25; First posted 2024-02-12 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Cervical Cancer; HPV Infection; Precancerous Lesion
Keywords: Prevention; Cervical cancer; HPV test; Self-sampling
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — HPV DNA smears from the cervix
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Not participating in screening: All women over 30 years of age who are not participating in screening or have not had a screening visit in less than 5 years.
  Interventions: Diagnostic Test: HPV DNA self-test
- Participating in the screening: All women over 30 years of age who regularly participate in screening but have not had an HPV test in the last 3 years.
  Interventions: Diagnostic Test: HPV DNA self-test

INTERVENTIONS:
Diagnostic Test: HPV DNA self-test — HPV DNA swab from the cervix performed by the patient herself.

SUMMARY:
One of the limitations of organized cervical screening in the Czech Republic is the lack of participation in preventive gynecological examinations. The aim of the project is to evaluate the benefits of self-sampling for HPV DNA in general practitioners' outpatient clinics to improve population participation in cervical screening.

DETAILED DESCRIPTION:
Organized cervical screening in the Czech Republic has a long-term participation rate of about 56% of the target population. Despite active invitations through health insurance companies, a part of the population is resistant and does not participate in screening visits to gynaecologists in the long term. A significant proportion of such women, however, regularly visit their general practitioner due to other comorbidities. The aim of the ASTRA project is to assess whether an effective way to increase the proportion of women attending cervical screening is to perform self-testing for HPV DNA in the GP's office.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent for statistical data processing and consent to the processing of personal data
* Age 30+
* HPV test never performed or performed more than 3 years ago or patient does not know

Exclusion Criteria:

* Refusal to participate
* Pregnancy and puerperium
* Menses
* History of hysterectomy
* HPV test performed <3 years ago with negative result
* Regular participation in screening and concurrent age 35, 45 or 55 years (test will be performed in the same year of screening).

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women over 30 years of age who meet the entry criteria for inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
To assess response rates to being approached about the possibility of self-testing for HPV in both study cohorts and overall. | Through study completion, an average of 1 year
  To compare the proportion of women who self-test for HPV DNA in a GP office versus those who refuse to take the test. To assess the overall proportion of women who self-test and the proportion in each study cohort.
Evaluation of the frequency of positivity of the HPV tests taken. | Through study completion, an average of 1 year
  Compare the proportion of women who will self-test positive for HPV DNA, including an assessment of positivity for HPV 16/18 and other HPV genotypes. To assess the overall proportion of women testing positive and the proportion in each study cohort.
Evaluation of follow-up gynaecological care in women who tested positive. | Through study completion, an average of 1 year
  To assess what proportion of women who self-test positive for HPV DNA will accept a gynecologic exam and to assess the results of the gynecologic visit.

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Cibulová, MS, Study Chair — Patient Organisation Veronica
Locations (2):
- Czechia (2):
  - CGOP, s.r.o., Prague
  - Department of Gynecology, Obstetrics and Neonatology, General University Hospital, First Faculty of Medicine, Charles University, Prague

IPD SHARING:
Plan to Share IPD: Undecided
All anonymised data will be available.

REFERENCES:
- [Background] Slama J, Dvorak V, Trnkova M, Skrivanek A, Hrabcova K, Ovesna P, Novackova M. Is phased implementation of HPV testing and triage with dual staining the way to transform organized cytology screening? Eur J Cancer Prev. 2024 Mar 1;33(2):168-176. doi: 10.1097/CEJ.0000000000000844. Epub 2023 Sep 21. PMID 37751376
- [Background] Sehnal B, Slama J. What next in cervical cancer screening? Ceska Gynekol. 2020 Winter;85(4):236-243. PMID 33562978
- [Background] Ngo O, Chloupkova R, Cibula D, Slama J, Mandelova L, Hejduk K, Hajduch M, Minka P, Koudelakova V, Jaworek H, Trnkova M, Vanek P, Dvorak V, Dusek L, Majek O. Direct mailing of HPV self-sampling kits to women aged 50-65 non-participating in cervical screening in the Czech Republic. Eur J Public Health. 2024 Apr 3;34(2):361-367. doi: 10.1093/eurpub/ckad229. PMID 38224266